CLINICAL TRIAL: NCT03245632
Title: Epidemiological Characteristics and Treatment Protocol for Carbapenem-Resistant Klebsiella Pneumoniae in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Prof., Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-CRKP
Record Dates: First submitted 2017-08-06; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Klebsiella Pneumoniae Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carbapenem-Resistant K. pneumoniae: Patients with clinical confirmed Carbapenem-Resistant Klebsiella pneumoniae infection.
  Interventions: Other: Carbapenem-Resistant Klebsiella pneumoniae
- Carbapenem-Sensitive K. pneumoniae: Any patients with clinical confirmed Carbapenem-Sensitive Klebsiella pneumoniae infection.

INTERVENTIONS:
Other: Carbapenem-Resistant Klebsiella pneumoniae — no intervention, this is an obervational study.
  Groups: Carbapenem-Resistant K. pneumoniae

SUMMARY:
Klebsiella pneumoniae is one of the most common pathogens causing nosocomial infection. Recently, the emergency of Carbapenem-Resistant Klebsiella pneumoniae (CRKP) had cause the clinical therapy be very difficult. However, there is not much empirical data as to the prevalence, risk factors, characteristics, and the rationality of the current therapy for the CRKP infection. Thus, the study was aimed to investigate the epidemiology and risk factors, characteristics, and the rationality of the current therapy for the CRKP infection.

DETAILED DESCRIPTION:
All the patients with culture positive of Klebsiella pneumoniae were screened and reported to the the clinical doctors and confirmed by them. And the clinical characteristics of the patiens, such as baseline data, outcomes etc, were recorded. Finially, to find the prevalence, risk factors, characteristics, and the rationality of the current therapy for the CRKP infection

ELIGIBILITY:
Inclusion Criteria:

* new confirmed noscomial infection of CRKP

Exclusion Criteria:

* Age<18, or >85 years old; Mixed infection of CRKP and other microbes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to all study hospitals and met the aboved eligibility
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
CRKP infection | 7 days
  Culture postitive results confirmed the infection of CRKP

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song YU, Doctor, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
For the time, we are not yet make determined to take the IPD plan